CLINICAL TRIAL: NCT01773694
Title: Impact of Early Post-Operative Water Exposure on Complications of Cutaneous Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: American Society for Dermatologic Surgery (Other)
Responsible Party: Principal Investigator, Todd V Cartee, Associate Professor of Dermatology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMC IRB 38335EP
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2020-09

CONDITIONS: Surgical Wound Infection
Keywords: Post-operative management; Post-operative complications; Post-operative treatment; water; skin; Dermatologic Surgical Procedures
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Water Exposure (Active Comparator): The Intervention group will receive written and verbal instructions to remove the dressing after 6 hours and wet the wound for at least 10 minutes. Wetting of the wound will include shower, tub bath, or pool exposure.
  Interventions: Behavioral: Early Water Exposure
- Standard Care (No Intervention): The Standard Care group will receive standard wound care instructions and verbal education by the staff to keep the dressing dry and intact for 48 hours.

INTERVENTIONS:
Behavioral: Early Water Exposure — The Early Water Exposure (Intervention) group will receive written and verbal instructions to remove the dressing after 6 hours and wet the wound for at least 10 minutes. Wetting of the wound will include shower, tub bath, or pool exposure.
  On subsequent days, all participants, regardless of group assignment, will wash the wound daily with soap and water, reapply white petrolatum and a dry dressing.
  Arms: Early Water Exposure

SUMMARY:
Patients are often counseled to keep a surgical wound dry for 2 to 3 days. The rationale is likely to decrease the risk of infection and bleeding. However, this has never been formally studied. Patient's routines are likely disrupted when they are asked to avoid wetting the area. The investigators will perform a controlled study to determine if avoidance of post-operative wetting is necessary.

DETAILED DESCRIPTION:
Physicians commonly instruct their patients to keep a wound dry for 2 to 3 days following surgery. The rationale may be that sources of water like a shower, bathtub, or swimming pool may increase the risk of infection. There may also be a concern that changing a dressing in the early post-operative period will increase the risk of bleeding complications. However, patient's routines and quality of life are disrupted when they are asked to avoid bathing, exercise, and swimming.

These issues have never been formally studied. This study will test the hypothesis of whether early post-operative wetting will have any influence on infection rates, bleeding complications, or the appearance of a surgical wound. Patients presenting to the Penn State Hershey dermatology clinic for the surgical removal of cancerous or non-cancerous skin lesions will be invited to participate. There will be no change to the standard surgical treatment. The dressing will be the same for all study participants. After surgery, study subjects who consent to participate will be randomized to receive one of two sets of post-operative instructions. One group will be directed to keep their initial post-operative dressing intact and dry for 48 hours. The second group will remove the dressing at 6 hours and wet the wound for 10 minutes in whatever manner they choose (shower, bath, pool, hot tub, etc.). After the initial dressing is removed (at 48 hours or 6 hours), both groups will perform identical post-operative care, consisting of cleansing the wound with soap and water followed by the application of petrolatum ointment and a dry dressing.

All participants will follow-up 7 to 14 days after surgery or earlier if they are experiencing any problems. At this time, the site will be assessed for clinical evidence of infection and bleeding. If the former is present, a bacterial culture will be obtained to confirm a wound infection and patients will be treated with an antibiotic. Physicians performing the assessment will be blinded to the patient's status (early wetting group or not). All subjects will also complete a questionnaire inquiring how and when they wet their wounds after surgery as well as two questionnaires asking how their quality-of-life and function were affected. Participants will again follow-up at 6 months when a blinded investigator will assess the cosmetic appearance of the scars using an established scar rating tool.

The data from this study will provide valuable evidence based guidance to surgeons in drafting wound care instructions for their patients. If the hypothesis proves correct, patients may be spared the inconvenience of post-operative water avoidance, diminishing the disruption to their lives caused by skin surgery.

ELIGIBILITY:
Inclusion Criteria:

1. subjects are capable of giving informed consent
2. patients undergoing any surgical treatment of benign and malignant lesions by any physician in the Dermatology department consisting of:

   1. standard excisional surgery or Mohs micrographic surgery with immediate reconstruction
   2. reconstruction with primary linear closure or adjacent tissue transfer with one or two layers of suture

Exclusion Criteria:

1. pregnancy
2. age younger than 18 years
3. will not be returning to the dermatology clinic in 7-14 days for suture removal
4. documented or suspected infection of the site prior to surgery
5. current treatment with systemic antibiotic therapy
6. staged excisions
7. delayed or staged reconstructions
8. wounds repaired with skin or cartilage grafts
9. management with secondary intention healing
10. surgical site on or near a mucosal surface where standard dressings are not typically used (eyelid, vermilion, etc.)
11. patients receiving prophylactic antibiotics
12. patients deemed on a case-by-case basis by their surgeon to have a high risk of post-operative bleeding and requiring prolonged application of a pressure dressing
13. history of skin sensitivity or reaction to white petrolatum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Post-operative wound infection | Post-operative day 7 to 14

SECONDARY OUTCOMES:
Incidence of post-operative bleeding complications | Post-operative day 7 to 14
Scar appearance | 6 months post-operatively (+-5 days)
  Using a non-invasive scoring tool, participants and a blinded physician will rate the appearance of the scar 6 months after the surgery.
Skin Specific Quality of Life | Post-operative days 7 to14
  Using a validated survey, information on the participants' quality of life will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Todd V Cartee, MD, Principal Investigator — Milton S. Hershey Medical Center; Joslyn S Kirby, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Department of Dermatology, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mudigonda T, Pearce DJ, Yentzer BA, Williford P, Feldman SR. The economic impact of non-melanoma skin cancer: a review. J Natl Compr Canc Netw. 2010 Aug;8(8):888-96. doi: 10.6004/jnccn.2010.0066. PMID 20870635
- [Background] Li J, Chen J, Kirsner R. Pathophysiology of acute wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):9-18. doi: 10.1016/j.clindermatol.2006.09.007. PMID 17276196
- [Background] Menke NB, Ward KR, Witten TM, Bonchev DG, Diegelmann RF. Impaired wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):19-25. doi: 10.1016/j.clindermatol.2006.12.005. PMID 17276197
- [Background] WINTER GD. Formation of the scab and the rate of epithelization of superficial wounds in the skin of the young domestic pig. Nature. 1962 Jan 20;193:293-4. doi: 10.1038/193293a0. No abstract available. PMID 14007593
- [Background] Ratz, J.L. Textbook of dermatologic surgery, (Lippincott-Raven, Philadelphia, 1998).
- [Background] Robinson, J.K. Surgery of the skin : procedural dermatology, (Elsevier Mosby, Philadelphia, 2005).
- [Background] Wolcott R, Dowd S. The role of biofilms: are we hitting the right target? Plast Reconstr Surg. 2011 Jan;127 Suppl 1:28S-35S. doi: 10.1097/PRS.0b013e3181fca244. PMID 21200270
- [Background] Smack DP, Harrington AC, Dunn C, Howard RS, Szkutnik AJ, Krivda SJ, Caldwell JB, James WD. Infection and allergy incidence in ambulatory surgery patients using white petrolatum vs bacitracin ointment. A randomized controlled trial. JAMA. 1996 Sep 25;276(12):972-7. PMID 8805732
- [Background] Chren MM, Lasek RJ, Flocke SA, Zyzanski SJ. Improved discriminative and evaluative capability of a refined version of Skindex, a quality-of-life instrument for patients with skin diseases. Arch Dermatol. 1997 Nov;133(11):1433-40. PMID 9371029
- [Background] Tsao S, Yao M, Tsao H, Henry FP, Zhao Y, Kochevar JJ, Redmond RW, Kochevar IE. Light-activated tissue bonding for excisional wound closure: a split-lesion clinical trial. Br J Dermatol. 2012 Mar;166(3):555-63. doi: 10.1111/j.1365-2133.2011.10710.x. Epub 2012 Jan 19. PMID 22032650
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848